CLINICAL TRIAL: NCT05453656
Title: Co-design, Development and Evaluation of the KIDNEY BEAM-KIDS Platform for Paediatric Kidney Transplant Recipients: a Feasibility Study
Brief Title: Development and Testing of the Kidney BEAM-KIDS Digital Platform for Children After Kidney Transplantation
Acronym: BEAM-KIDs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Margaret University (Other)
Collaborators: Sheffield Hallam University (Other); King's College Hospital NHS Trust (Other); Keele University (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Glasgow Royal Hospital for children (Unknown)
Responsible Party: Principal Investigator, Pelagia Koufaki, PhD, Reader, Exercise Physiology and Rehabilitation Sciences, Queen Margaret University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P2008QMU
Record Dates: First submitted 2022-06-20; First posted 2022-07-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Kidney Transplantation
Keywords: exercise; child; adolescent; quality of life
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise (Other): live and on demand exercise sessions on the Kidney BEAM-KIDS platform
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — physical activity promotion and engagement following kidney transplantation
  Other Names: kidney transplantation

SUMMARY:
Children and young people (CYP) with chronic kidney disease (CKD) say that physical activity, school, social activities and tiredness are the main issues they want to improve. Kidney-BEAM, a digital health platform designed for adults with CKD, provides a combination of live and on-demand exercise classes to encourage physical activity and movement but is currently not available to CYP with CKD. Therefore, investigators will work with CYP with CKD, parents/carers and healthcare professionals to find out if a CYP-related version (Kidney BEAM-KIDS), could be developed to encourage exercise options that are enjoyable, safe and sustainable. In this project, CYP who have received a KT will be invited by their local clinical teams to try out Kidney BEAM-KIDS; this will include exercise-based classes delivered in age-appropriate groups where CYP will be able to get peer support. Kidney BEAM-KIDS will include features to help motivation such as badges and celebrations when reaching targets. The CYP will be asked to participate in discussions and complete several questionnaires at three time-points over 12 months to explore how CYP feel about themselves and aspects of their lives such as friendships and school, how physically active they are, their preferred types of foods, activities they do, and their health. This will help the investigators a) understand how acceptable Kidney BEAM-KIDS is to CYP, b) determine whether it needs any changes/improvements, and c) identify key issues around how best to gather data and answer research questions about physical activity benefits in CYP with CKD.

DETAILED DESCRIPTION:
Kidney transplantation (KT) is the preferred and most prevalent treatment in CYP with CKD but is associated with increased risk of cardiovascular complications, insulin resistance, and diabetes, with likely contributors being visceral obesity and low lean body mass. In general paediatric populations, all of the above are favourably modified by regular/varied PA. The benefits and risks of PA for CYP with CKD are, however, less well established and available data are mainly from cross-sectional studies. Kidney-BEAM is a digital health platform for adults with CKD, which provides live and on-demand exercise classes. The investigators propose to adapt the kidney BEAM platform to kidney BEAM-KIDS for CYP with CKD to access activities adapted to their needs and document benefits on outcomes that matter to them.

Aims and methods: A single-arm, multi-centre, feasibility study, with a mixed-method design using an effectiveness and theory-based perspective. Investigators will examine the feasibility and acceptability of (a) Kidney BEAM-KIDS as the intervention and delivery setting in CYP following KT, and (b) the evaluation design for addressing all recommended core elements (context, engaging stakeholders, identifying key uncertainties, refining the intervention, economic considerations) to inform the development of a clinical evaluation trial The team will aim to recruit about 30 participants between 6-17 years of age. Research questions:

1. What are participants' experiences of Kidney BEAM-KIDS and views on its feasibility, acceptability and benefits?
2. What type and quantity of adverse events (if any) are experienced over an observation period of 7-12 months?
3. What are the study recruitment and retention rates?
4. What is the acceptability of data collection methods and rate of outcome measure completion?
5. What are the variability and patterns of change in outcomes to determine a primary outcome measure and calculate sample size for a future study?
6. What is the feasibility of a future health economic evaluation?

Outcomes: Quantitive data: demographic, clinical and physical characteristics, adverse events and hospitalisations, 4-7 day dietary intake diaries, at 3 time points: before and after KT and after 12 weeks exposure to Kidney BEAM-KIDS. Selection of outcomes was based on i) the potential impact on outcomes that matter to CYP (multidimensional PedsQLv4, self perception profile, Physical activity questionnaire, BEAM-KIDS platform use metrics), (ii) participants' wide age range (6-17 years), and iii) the need to minimise face-to-face assessments where possible due to the wide geographical spread of recruiting centres. Physical function outcomes (strength and cardiorespitatory fitness) will be collected in person if possible. Qualitative data: via remote semi-structured individual interviews and focus groups using a process evaluation approach to explore experiences, attitudes, preferences, suggestions to inform future directions.

ELIGIBILITY:
Inclusion Criteria:

* CYP of school age between 6 and 17 years attending a paediatric transplant centre
* Likely to require a KT within 12 months
* No intended date of transition to adult services within 12 months

Exclusion Criteria:

* Inability or absolute contraindications to engaging in PA
* Severe bone disease
* Cancer/leukaemia or HIV treatment within the 12 months before enrolment
* Enrolment in other clinical trials in which treatment is masked.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — self reported
Enrollment: 30 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life score | change from baseline to 12 and 24 weeks post kidney transplantation and exercise
  the multidimensional PedsQLv4 questionnaire and relevant sub-module questionnaires on fatigue and transplantation will be used to estimate scores that reflect the domains of physical functioning, emotional functioning, social functioning, school functioning, general fatigue, sleep/rest fatigue and cognitive fatigue, treatment anxiety

SECONDARY OUTCOMES:
Frequency and type of physical activity | change from baseline to 12 and 24 weeks post kidney transplantation and exercise
  the self-reported Physical Activity Questionnaire - PAQ for CYP will be used to capture data on PA patterns
type and quantity of food groups consumed | change from baseline to 12 and 24 weeks post kidney transplantation and exercise
  4-7 day diaries will be used to capture and analyse nutritional intake information
adverse events | change from baseline to 12 and 24 weeks post kidney transplantation and exercise
  episodes of hospitalisations and other infection events will be captured via medical records
kidney BEAM-KIDS platform metrics | change from 12 weeks post kidney transplantation to 12 weeks post exercise
  minutes spent on physical activity and engagement with the digital health platform
qualitative exploration of trial acceptability and participant experience | at 12 weeks post kidney transplantation
  focus groups and semi structured interviews with participants and families will be used to capture qualitative data
qualitative exploration of trial acceptability and participant experience | at 12 weeks post exercise
  focus groups and semi structured interviews with participants and families will be used to capture qualitative data

CONTACTS AND LOCATIONS:
Locations (1):
- Glasgow Royal Hospital for Children, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan yet